CLINICAL TRIAL: NCT04014738
Title: The Prognostic Value of Human Papilloma Virus in Nasopharyngeal Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Other Study IDs: 0190-19-RMB-CTIL
Record Dates: First submitted 2019-07-09; First posted 2019-07-10 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Histopathological slides
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
It is well established that HPV infection has a casual and is a prognostic factor in several cancer types, including oropharynx. We wish to examine if HPV infection has a prognostic significance in nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* nasopharyngeal carcinoma patients treated in our institute between 2008-2018

Exclusion Criteria:

* missing clinical data
* 2nd Head and neck primary cancer
* very locally advanced or distant metastatic nasopharyngeal carcinoma
* Prior radiation therapy to the head and neck region

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with nasopharyngeal carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-07-20 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Eran S Fridman, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam medical center, Haifa, Israel